CLINICAL TRIAL: NCT04483843
Title: Impact of Cosmic Weather on Pre-hospital Incidence of Cardiogenic Pulmonary Edema
Brief Title: Cosmic Weather and Cardiogenic Pulmonary Edema
Status: Completed | Type: Observational
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other); Institute of Experimental Physics, Slovak Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: 2019-03
Record Dates: First submitted 2019-08-03; First posted 2020-07-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Edema Cardiac Cause
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPE patients: All patients prehospitally treated for cardiogenic pulmonary edema in the pre-hospital emergency setting in the Central Bohemian region, Czech Republic.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be performed while it is retrospective observational study.

SUMMARY:
Retrospective clinical study to evaluate whether there is any correlation between the pre-hospital incidence of cardiogenic pulmonary oedema (CPE) in the selected region and the space weather parameters.

DETAILED DESCRIPTION:
Emergency Medical Service of the Central Bohemian Region is the exclusive provider of primary pre-hospital emergency care in the Central Bohemian Region, Czech Republic. The region includes both the rural and urban population, in total of 1 315 299 inhabitants on a total area of 11 015 km2. A computer search of patients with dyspnoea between 1.10.2008 and 30.6.2014 will be conducted and all cases of cardiogenic pulmonary oedema will be selected.

Physical parameters of space weather and geomagnetic field disturbances will be obtained from the database of Institute of Experimental Physics, Slovak Academy of Sciences, Slovak Republic. The datasets will be analysed whether there is any correlation between the pre-hospital incidence of CPE in the selected region and the parameters of space weather and geomagnetic field disturbances.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated by Emergency Medical Service of the Central Bohemian Region for cardiogenic pulmonary edema between 1.10.2008 and 30.6.2014.

Exclusion Criteria:

* Dyspnea from other cause than cardiogenic pulmonary edema.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from the registry of the Emergency Medical Service of the Central Bohemian Region, Czech Republic who were treated prehospitally for cardiogenic pulmonary edema between 1.10.2008 and 30.6.2014.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Significant correlation between incidence of CPE and activity of the space weather | 4 years
  Significant correlation between incidence of CPE and activity of the space weather
Significant correlation between incidence of CPE and the degree of the geomagnetic field disturbance | 4 years
  Significant correlation between incidence of CPE and the degree of the geomagnetic field disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Emergency Medical Service of the Central Bohemian Region, Czech Republic
Locations (1):
- Emergency Medical Service of the Central Bohemian Region, Beroun, Central Bohemia, Czechia

IPD SHARING:
Plan to Share IPD: No
No sharing anticipated.